CLINICAL TRIAL: NCT00448474
Title: Mail-Delivered Arthritis Self-Management Education -- Years 1, 2, Carryover
Brief Title: Development and Evaluation of A Mailed Arthritis Self-Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina (Other)
Collaborators: Stanford University (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 05-1163-1-3
Record Dates: First submitted 2007-03-14; First posted 2007-03-16 (Estimated); Last update posted 2007-03-16 (Estimated); Status verified 2007-03

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis
Keywords: Disease self-management; Community program
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Mailed Arthritis Self-Management Education

SUMMARY:
The purpose of this study is twofold, to develop and test the effectiveness of a mailed arthritis self-management education intervention.

DETAILED DESCRIPTION:
Effective self-management education programs for persons with arthritis have been developed, delivered in various formats, and found effective. Because of limited resources, however, many state health departments have found dissemination difficult, particularly to vulnerable populations. Researchers at the University of North Carolina at Chapel Hill and Stanford University will develop an evidence-based mail-delivered arthritis self-management program (Arthritis Yes I Can) that is feasible for state health department use and that can be self-tailored to meet the needs of diverse populations. The study will be conducted in three phases.

During Phase One (Development) researchers will collaborate with CDC advisors, arthritis experts from state health departments, and Project consultants to develop the curriculum and compact disc (CD) and print materials for mail-delivery. We will base Arthritis Yes I Can on curricula of two evidence-based programs, the Arthritis Self Help Course (ASHC) and the Chronic Disease Self Management Program (CDSMP), and develop English and Spanish versions.

During Phase Two (Evaluation) we will utilize both a randomized pre-test post-test (four month) delayed treatment control group design and a longitudinal cohort design to evaluate program effectiveness. We will recruit 900 individuals, 300 African Americans, 300 other English speakers, and 300 Spanish speakers, who: 1. Have been diagnosed with osteoarthritis or rheumatoid arthritis, or meet CDC criteria for chronic joint symptoms; 2. Are at least 18 years of age; and 3. Are able to complete informed consent, enrollment forms, and interviews/questionnaires. In addition, participants must not have participated in a previous arthritis self-management program and have access to a CD player. They must be willing to commit 8-12 hours of self-study over 4-6 weeks. We will use multiple recruitment methods, emphasizing collaboration with state and local health departments. We will measure: 1. Knowledge of Arthritis and Arthritis Self-Management, 2. Health-related Quality of Life (Self-reported Health, Pain, Disability, Fatigue, Activity Limitation, Health Distress, and Depression); 3. Health Care Utilization; 4. Self-Management Behaviors; and 5. Self-Efficacy for Arthritis Self-Management and Arthritis Helplessness. We will also evaluate participant satisfaction with mail delivery, and determine the relative success of all recruitment efforts.

If the intervention is found effective in Phase Two, we will offer guidance to the Arthritis Program of the Centers for Disease Control and Prevention in adopting and distributing Arthritis Yes I Can (Phase Three, Dissemination).

ELIGIBILITY:
Inclusion Criteria:

* Report MD diagnosis of osteoarthritis or rheumatoid arthritis, or meet CDC criteria for chronic joint symptoms
* Are at least 18 years of age
* Are able to complete informed consent, enrollment forms, and interviews/questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900
Dates: Start 2005-11; Study Completion 2006-07

PRIMARY OUTCOMES:
Health-related Quality of Life (Self-reported Health, Pain, Disability, Fatigue, Activity Limitation, Health Distress)
Health Care Utilization
Self-Management Behaviors
Self-Efficacy for Arthritis Self-Management

CONTACTS AND LOCATIONS:
Overall Officials: Jean Goeppinger, PhD, BSN, Principal Investigator — University of North Carolina, Chapel Hill; Kate Lorig, DrPH, BSN, Principal Investigator — Stanford University
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States